CLINICAL TRIAL: NCT03956108
Title: Active Surveillance for Low-risk Prostate Cancer - Evaluation of the Efficacy of Minimally Invasive Active Surveillance
Acronym: STHLM3AS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Anna Lantz, Principal Investigator, Karolinska Institutet
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018/276-31/2
Record Dates: First submitted 2019-05-15; First posted 2019-05-20 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Prostate Cancer
Keywords: Active Surveillance
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MRI/Fusion biopsies (Experimental): Stockholm3+MRI+targeted biopsies
  Interventions: Diagnostic Test: MRI+targeted biopsies+Stockholm3-test
- Systematic biopsies (Active Comparator): PSA+systematic biopsies
  Interventions: Diagnostic Test: PSA + systematic biopsies

INTERVENTIONS:
Diagnostic Test: MRI+targeted biopsies+Stockholm3-test — MRI, evaluation in accordance with PI-RADS v2, and targeted biopsies. Stockholm3-test.
  Arms: MRI/Fusion biopsies
Diagnostic Test: PSA + systematic biopsies — Systematic biopsies and PSA test
  Arms: Systematic biopsies

SUMMARY:
The STHLM3-AS study will evaluate the specificity of a new proposed protocol for active surveillance using the Stockholm3 test in combination with MRI targeted biopsies for prostate cancer detection in men with diagnosed low-risk prostate cancer undergoing active surveillance in comparison to conventional follow up using PSA and systematic biopsies.

DETAILED DESCRIPTION:
The study design is a cross-sectional study, using a paired design, evaluating our proposed protocol (Stockholm3+MRI+targeted biopsies) versus the standard protocol (PSA+systematic biopsies).

Men from the STHLM3 study, diagnosed with low risk prostate cancer and currently on AS will be invited to the study. Eligible individuals have to be alive without any severe comorbidity and without a history of initiating treatment; surgery, radiation, hormone therapy or chemotherapy. To avoid the need for additional biopsies, invitation will be synchronized with timing for planned follow-up within the AS program for each individual.

At baseline blood will be drawn for PSA and Stockholm3 analyses. The patient will be asked to fill out a study specific questionnaire with questions on anxiety and quality of life. Additionally, a bi-parametric MRI evaluated in line with PI-RADS v2 guidelines will be performed. For men with PIRADS ≥ 3 targeted and systematic biopsies will be performed. For men with PIRADS<3 only systematic biopsies will be performed.

Main outcome measurement will be number of detected significant cancers by each method. Further outcome measurements are the number of performed prostate biopsies with each method and level of anxiety and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Men in the STHLM3 study, diagnosed with a low risk prostate cancer and on AS

Exclusion Criteria:

* History of treatment for prostate cancer; surgery, radiation, chemotherapy or hormonal treatment.
* Severe illnesses such as metastatic cancers, severe cardio-vascular disease or dementia
* Contraindications for magnetic resonance imaging (MRI) e.g. pacemaker, magnetic cerebral clips, cochlear implants or severe claustrophobia.

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only men present with prostate cancer
Enrollment: 280 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Specificity of minimally invasive active surveillance | Up to five years
  Number of biopsies using the Stockholm3 test in combination with MRI/targeted biopsies vs. number of systematic biopsies at equal sensitivity for detecting Gleason Score ≥ 7 disease

SECONDARY OUTCOMES:
Predictive value of Stockholm3 test velocity | Up to five years
  Stockholm3 test velocity
Clinically significant cut off for Stockholm3 test as a monitoring test | Up to five years
  Stockholm3 test cutoff (0-100% risk)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Lantz, MD PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Solna, Sweden

IPD SHARING:
Plan to Share IPD: No
Information obtained in the study will be collected in one database. The purpose of the database is to collect study data in a proper and safe way for a long time. All information about the participants will be treated with utmost confidentiality and with strong safeguards to preserve their anonymity. Information that can be used to identify the participant (such as name, address and social security numbers) is always kept separate from other data (such as survey responses and blood tests). All questionnaire data and test results will be treated to prevent unauthorized access to them. The samples will get a unique code so that outsiders cannot identify them. The participants' samples are treated in accordance with the Swedish Biobank Act.
  Everyone who works with STHLM3 are under confidentiality agreements. Results from the study are presented only as statistics in which individual answers cannot be traced.

DOCUMENTS (1):
  • Informed Consent Form (2019-05-31): https://cdn.clinicaltrials.gov/large-docs/08/NCT03956108/ICF_000.pdf